CLINICAL TRIAL: NCT03098394
Title: Use of a Rapid Turnaround Test for Gonorrhea & Chlamydia to Improve Treatment of Women Presenting With Possible Sexually Transmitted Infections
Brief Title: Use of a Rapid Test for Gonorrhea & Chlamydia for Women Presenting With Possible Sexually Transmitted Infections
Status: Terminated | Phase: Not Applicable | Type: Interventional
Why Stopped: Low enrollment
Sponsor: University of Maryland, Baltimore (Other)
Responsible Party: Principal Investigator, Richard Gentry Wilkerson, Assistant Professor, University of Maryland, Baltimore
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Diagnostic
Other Study IDs: HP-00072766
Record Dates: First submitted 2017-03-27; First posted 2017-03-31 (Actual); Results first posted 2023-08-31 (Actual); Last update posted 2023-08-31 (Actual); Status verified 2023-08

CONDITIONS: Sexually Transmitted Infection; Gonorrhea Female; Chlamydia Females
Keywords: Rapid turnaround test; RTAT; Gonorrhea; Chlamydia; STI
MeSH Terms: conditions — Sexually Transmitted Diseases; Gonorrhea; Chlamydia Infections | interventions — Polymerase Chain Reaction

STUDY DESIGN:
Intervention Model Description: This is a prospective, non-blinded, randomized clinical control trial
Who Masked: Participant, Care Provider, Investigator
Masking Description: Participants, investigators, and care providers will be masked to the experimental or control arm prior to enrollment in the study. Once the participant has been enrolled in the study, they will be randomized to either the control arm or the experimental arm. Once randomization has occurred, participants, care providers, and the investigators will know which group the participants are in.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: Yes | US Export: Yes

ARMS (2):
- Rapid Turnaround Test (Experimental): Patients randomized to this arm will be tested for a sexually transmitted infection (STI) with both the rapid nucleic acid amplification test (NAAT) as well as the conventional polymerase chain reaction (PCR) test. The results from the rapid turnaround test will guide providers on treatment decisions for a possible STI. The results from the PCR test will be used to verify the results of the rapid turnaround test.
  Interventions: Device: Cepheid Xpert CT/NG Rapid Turnaround Test; Device: Polymerase chain reaction (PCR)
- Usual Care (Active Comparator): Patients randomized to this arm will be tested for a sexually transmitted infection (STI) using the conventional PCR test. The results from the PCR test normally take approximately 48-72 hours and these patients will likely receive treatment based on the decision of the clinical provider. The results from the PCR test will be used to verify the decision of the clinical provider to treat or withhold treatment for a possible STI.
  Interventions: Device: Polymerase chain reaction (PCR)

INTERVENTIONS:
Device: Cepheid Xpert CT/NG Rapid Turnaround Test — This diagnostic test will be used to help clinicians determine the need for antibiotic prescriptions in patients with a suspected sexually tract infection.
  Other Names: GeneXpert
  Arms: Rapid Turnaround Test
Device: Polymerase chain reaction (PCR) — This is the standard of care for diagnosis of a suspected sexually transmitted infection.
  Other Names: PCR

SUMMARY:
The purpose of this study is to evaluate the effect of utilizing a rapid turnaround CT/NG test on treatment of female patients in the emergency department or urgent care setting with possible STIs.

DETAILED DESCRIPTION:
All females ages 18-55 presenting to the University of Maryland Medical Center Emergency Department or Urgent Care whose provider suspects sexually transmitted infection will be offered study enrollment and be randomly assigned to either the control or the experimental group. Both groups will have a urinalysis, a pregnancy test, a pelvic exam, and an endocervical sample collected, but the experimental group's urine will be used to run the rapid turnaround test (RTAT) instead of the standard PCR. Data will be collected regarding provider decision making, length of stay in the emergency department, patient satisfaction, clinician satisfaction, further healthcare sought by patient, and cost surrounding each treatment.

ELIGIBILITY:
Inclusion Criteria:

* Female patients age 18-55
* Signs or symptoms consistent with sexually transmitted infection
* Medical provider willing to consider the result of the rapid turnaround test in decision to treat for gonorrhea/chlamydia
* Must have a urine specimen obtained and a pelvic exam performed as part of the anticipated standard of care evaluation
* Provides informed consent

Exclusion Criteria:

* Signs of systemic infection
* Patient in whom the provider is unwilling to consider the result of the rapid turnaround test
* Patient who reports being treated for either gonorrhea or chlamydia in the preceding 3 months
* Patients undergoing evaluation for sexual assault
* Patients that are known to be pregnant or express concern that they may be pregnant
* Incarcerated patients
* Students/Employees of the facility
* Presence of any other condition(s) that the investigator feels makes the patient unsuitable for study inclusion.

Ages: 18 Years to 65 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Gender Based: Yes — Participant eligibility is not based on self-representation of gender identity. All participants in this study will receive a pelvic exam in the emergency department as well as a cervical swab for diagnostic testing.
Enrollment: 64 (Actual)
Dates: Start 2018-09-24 (Actual); Primary Completion 2022-03-25 (Actual); Study Completion 2023-06-20 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Richard G Wilkerson, MD, Principal Investigator — University of Maryland, Baltimore
Locations (1):
- University of Maryland Medical Systems, Baltimore, Maryland, United States

IPD SHARING:
Plan to Share IPD: No
We do not plan on sharing any individual participant data with other researchers

REFERENCES:
- [Background] Brook G. The performance of non-NAAT point-of-care (POC) tests and rapid NAAT tests for chlamydia and gonorrhoea infections. An assessment of currently available assays. Sex Transm Infect. 2015 Dec;91(8):539-44. doi: 10.1136/sextrans-2014-051997. Epub 2015 May 2. PMID 25935930
- [Background] Gaydos CA. Review of use of a new rapid real-time PCR, the Cepheid GeneXpert(R) (Xpert) CT/NG assay, for Chlamydia trachomatis and Neisseria gonorrhoeae: results for patients while in a clinical setting. Expert Rev Mol Diagn. 2014 Mar;14(2):135-7. doi: 10.1586/14737159.2014.871495. Epub 2014 Jan 23. PMID 24450867
- [Background] Gaydos CA, Van Der Pol B, Jett-Goheen M, Barnes M, Quinn N, Clark C, Daniel GE, Dixon PB, Hook EW 3rd; CT/NG Study Group. Performance of the Cepheid CT/NG Xpert Rapid PCR Test for Detection of Chlamydia trachomatis and Neisseria gonorrhoeae. J Clin Microbiol. 2013 Jun;51(6):1666-72. doi: 10.1128/JCM.03461-12. Epub 2013 Mar 6. PMID 23467600
- [Background] Holley CE, Van Pham T, Mezzadra HM, Willis GC, Witting MD. Overtreatment of gonorrhea and chlamydial infections in 2 inner-city emergency departments. Am J Emerg Med. 2015 Sep;33(9):1265-8. doi: 10.1016/j.ajem.2015.06.009. Epub 2015 Jun 12. PMID 26119905
- [Background] Newman LM, Moran JS, Workowski KA. Update on the management of gonorrhea in adults in the United States. Clin Infect Dis. 2007 Apr 1;44 Suppl 3:S84-101. doi: 10.1086/511422. PMID 17342672
- [Background] Tabrizi SN, Unemo M, Golparian D, Twin J, Limnios AE, Lahra M, Guy R; TTANGO Investigators. Analytical evaluation of GeneXpert CT/NG, the first genetic point-of-care assay for simultaneous detection of Neisseria gonorrhoeae and Chlamydia trachomatis. J Clin Microbiol. 2013 Jun;51(6):1945-7. doi: 10.1128/JCM.00806-13. Epub 2013 Apr 3. PMID 23554203

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | Rapid Turnaround Test | Usual Care
Started | 30 | 34
Completed | 30 | 33
Not Completed | 0 | 1
Not completed — Pregnancy | 0 | 1

BASELINE CHARACTERISTICS:
Population: All analyzed patients included
Groups:
- Total: Total of all reporting groups
Arm/Group | Rapid Turnaround Test | Usual Care | Total
Number analyzed (Participants) | 30 | 33 | 63
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0
  Between 18 and 65 years | 30 | 33 | 63
  >=65 years | 0 | 0 | 0
Age, Continuous [Mean (Full Range); unit: years] | 30.3 [18 to 55] | 29 [19 to 50] | 29.6 [18 to 55]
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 30 | 33 | 63
  Male | 0 | 0 | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0
  Asian | 0 | 0 | 0
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0
  Black or African American | 0 | 0 | 0
  White | 0 | 0 | 0
  More than one race | 0 | 0 | 0
  Unknown or Not Reported | 30 | 33 | 63
Region of Enrollment [Number; unit: participants]
  United States | 30 | 33 | 63
Presence of signs or symptoms of STIs [Count of Participants; unit: Participants] | 30 | 33 | 63

OUTCOME MEASURES:

1. Primary Outcome: Number of Participants Treated With Antibiotics
Description: Evaluate the effect of a rapid turnaround CT/NG test compared to standard of care on antibiotic prescription for female patients with STI.
Time Frame: 7 days
Population: Intention to treat
Measure: Count of Participants; unit: Participants
Arm/Group | Rapid Turnaround Test | Usual Care
Number analyzed (Participants) | 30 | 33
Participants | 4 | 10

2. Secondary Outcome: Length of Stay (Minutes)
Description: Evaluate the effect of utilizing a rapid turnaround CT/NG test on length of stay (minutes) in the Emergency Department.
Time Frame: 7 days
Measure: Mean (Standard Deviation); unit: minutes
Groups:
- Rapid Turnaround Test: Subjects who received the RTAT
- Usual Care: Subjects who were assigned to the usual care group only
Arm/Group | Rapid Turnaround Test | Usual Care
Number analyzed (Participants) | 30 | 33
minutes | 200.6896552 (48.12936692) | 129.6060606 (60.9717862)

3. Secondary Outcome: Percentage of Patients With Rapid Turnaround CT/NG (RPAT) Tests That Are CONSISTENT With Usual Care Test (PCR) in Subjects That Had Both Performed.
Description: Compare the congruence of test results between the rapid turnaround CT/NG test with the usual care test (send out PCR) in subjects that have both performed (Experimental Group).
Time Frame: 7 days
Population: Four patients received indeterminate results on either their RTAT or their Usual Care (PCR) tests.
Measure: Number; unit: percentage of total RTAT + PCR patients
Groups:
- Subjects Who Received Both RTAT and Usual Care Tests: Subjects who received RTAT and Usual Care Tests (PCR) AND received official (non-indeterminate) test results.
Arm/Group | Subjects Who Received Both RTAT and Usual Care Tests
Number analyzed (Participants) | 26
percentage of total RTAT + PCR patients | 92.307

4. Secondary Outcome: Healthcare Costs.
Description: Evaluate the effect of utilizing a rapid PCR test on healthcare costs.
Time Frame: 7 days
Population: Heatlhcare cost data was not collected, thus could not be analyzed and reported.
Arm/Group | Rapid Turnaround Test | Usual Care
Number analyzed (Participants) | 0 | 0

5. Secondary Outcome: Average Score for Patient Satisfaction With Provider Explanation.
Description: Evaluate patient satisfaction with provider's explanations for the 2 diagnostic groups. Patients were asked to rate their satisfaction with their provider's explanations on a five point scale, with 0 being "not at all satisfied" and 4 being "very satisfied."
Time Frame: 7 days
Population: Patient counts for average satisfaction with provider explanation differ from total patient counts due to difficulty contacting patients for satisfaction surveys.
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Rapid Turnaround Test | Usual Care
Number analyzed (Participants) | 26 | 30
score on a scale | 3.346153846 (0.745241314) | 3.24137931 (0.872401137)

6. Secondary Outcome: Average Score for Patient Satisfaction With Treatment Effectiveness.
Description: Evaluate patient satisfaction with treatment effectiveness for the 2 diagnostic groups. Patients were asked to rate their satisfaction with their treatment effectiveness on a five point scale, with 0 being "not at all satisfied" and 4 being "very satisfied."
Time Frame: 7 days
Population: Patient counts for average satisfaction with treatment effectiveness differ from total patient counts due to difficulty contacting patients for satisfaction surveys.
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Rapid Turnaround Test | Usual Care
Number analyzed (Participants) | 26 | 30
score on a scale | 3.153846154 (0.731699812) | 3.206896552 (0.726012118)

7. Secondary Outcome: Average Score for Patient Satisfaction With Overall Experience.
Description: Evaluate patient satisfaction with overall experience during visit for the 2 diagnostic groups. Patients were asked to rate their satisfaction with their wait times on a five point scale, with 0 being "not at all satisfied" and 4 being "very satisfied."
Time Frame: 7 days
Population: Patient counts for average satisfaction with overall experience differ from total patient counts due to difficulty contacting patients for satisfaction surveys.
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Rapid Turnaround Test | Usual Care
Number analyzed (Participants) | 26 | 30
score on a scale | 3.346153846 (0.561591146) | 3.275862069 (0.797162455)

8. Secondary Outcome: Number of Patients That Required Follow-up Care Within 7 Days
Description: Compare need for additional healthcare utilization between the groups.
Time Frame: 7 days
Population: Total number of participants for this analysis differ from total number of participants in overall study due to difficulty contacting some patients for data collection after initial hospital visit.
Measure: Count of Participants; unit: Participants
Arm/Group | Rapid Turnaround Test | Usual Care
Number analyzed (Participants) | 27 | 30
Participants | 4 | 1

9. Secondary Outcome: Average Score for Patient Satisfaction With Wait Times During Visit.
Description: Evaluate patient satisfaction with wait times during visit for the 2 diagnostic groups. Patients were asked to rate their satisfaction with their wait times on a five point scale, with 0 being "not at all satisfied" and 4 being "very satisfied."
Time Frame: 7 days
Population: Patient counts for average satisfaction with wait times differ from total patient counts due to difficulty contacting patients for satisfaction surveys.
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Rapid Turnaround Test | Usual Care
Number analyzed (Participants) | 26 | 30
score on a scale | 3.038461538 (0.999230473) | 2.931034483 (0.923155864)

ADVERSE EVENTS:
Time Frame: 7 Days
Arm/Group | Rapid Turnaround Test | Usual Care
All-Cause Mortality (participants affected / at risk) | 0/30 | 0/33
Serious Adverse Events (participants affected / at risk) | 0/30 | 0/33
Other Adverse Events (participants affected / at risk) | 0/30 | 0/33

LIMITATIONS AND CAVEATS:
Early termination leading to small numbers of subjects enrolled

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No

DOCUMENTS (1):
  • Study Protocol (2018-07-02): https://cdn.clinicaltrials.gov/large-docs/94/NCT03098394/Prot_001.pdf